CLINICAL TRIAL: NCT01194570
Title: A Phase III, Multicentre, Randomized, Parallel-group, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ocrelizumab in Adults With Primary Progressive Multiple Sclerosis
Brief Title: A Study of Ocrelizumab in Participants With Primary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA25046; 2010-020338-25 (EudraCT Number)
Record Dates: First submitted 2010-08-28; First posted 2010-09-03 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Participants with primary progressive multiple sclerosis (PPMS) received placebo matched to ocrelizumab at a schedule interval of 24 weeks up to at least 120 weeks.
  Interventions: Drug: Ocrelizumab; Other: Placebo
- Ocrelizumab 600 mg (Placebo Comparator): Participants with PPMS received ocrelizumab as two IV infusions of 300 mg separated by 14 days at a scheduled interval of every 24 weeks up to at least 120 weeks.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Two IV infusions of 300 mg in each treatment cycle of double blind treatment period; two IV infusions of ocrelizumab 300 mg for Cycle 1 and single IV infusion of ocrelizumab 600 mg for subsequent cycles in OLE phase.
Other: Placebo — Two IV infusions of placebo matched to ocrelizumab in each treatment cycle of double blind treatment period.
  Arms: Placebo

SUMMARY:
This randomized, parallel group, double-blind, placebo controlled study will evaluate the efficacy and safety of ocrelizumab in participants with primary progressive multiple sclerosis. Eligible participants will be randomized 2 : 1 to receive either ocrelizumab or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary progressive multiple sclerosis (according to revised McDonald criteria)
* EDSS at screening from 3 to 6.5 points
* Disease duration from onset of MS symptoms less than (<) 15 years if EDSS greater than (>) 5.0; <10 years if EDSS greater than or equal to (>/=) 5.0
* Sexually active male and female participants of reproductive potential must use two methods of contraception throughout the study treatment phase and for 48 weeks after the last dose

Exclusion Criteria:

* History of relapsing remitting MS, secondary progressive, or progressive relapsing MS at screening
* Inability to complete an MRI (contraindications for MRI)
* Known presence of other neurologic disorders
* Known active infection or history of or presence of recurrent or chronic infection
* History of cancer, including solid tumors and hematological malignancies (except for basal cell, in situ squamous cell carcinomas of the skin and in situ carcinoma of the cervix that have been excised and resolved)
* Previous treatment with B-cell targeted therapies (e.g. rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
* Any previous treatment with lymphocyte trafficking blockers, with alemtuzumab, anti-cluster of differentiation 4 (CD4), cladribine, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 735 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2015-07-23 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (184):
- United States (37):
  - Phoenix Neurological Associates Ltd, Phoenix, Arizona
  - Barrow Neurology Clinic, Phoenix, Arizona
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - Arizona Neuroscience Research LLC, Phoenix, Arkansas
  - Sutter East Bay Medical Foundation, Berkeley, California
  - MS Center of Southern California, Newport Beach, California
  - Univ of CA Davis Med Ctr; Neurology, Sacramento, California
  - Univ of CA San Francisco; Department of Neurology, San Francisco, California
  - University of Colorado; Anschutz Medical Campus Department of Neurology, Aurora, Colorado
  - University of Miami School of Medicine; Dept. of Neurology Movement Disorder Center, Miami, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Prairie Village, Kansas
  - Wayne State University; Department of Neurology, Detroit, Michigan
  - Henry Ford Health System; Neurology & Neurosurgery, Detroit, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - University of Minnesota; Clin. Neuro Research Unit, Minneapolis, Minnesota
  - Washington University School of Medicine; Department of Neurology, St Louis, Missouri
  - Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico; MS Specialty Clinic, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - Weill Medical College of Cornell University; Judith Jaffe MS Ctr, New York, New York
  - Mount Sinai School of Medicine; Neurology, New York, New York
  - Comprehensive MS Care Center at South Shore Neurologic Assoc., Patchogue, New York
  - Neurology Assoc of Stony Brook, Stony Brook, New York
  - Carolinas Medical Center; Ms Center, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - The Ohio State University Wexner Medical Center; Department of Neurology, Columbus, Ohio
  - Oklahoma Medical Research Foundation; MS Center of Excellence, Oklahoma City, Oklahoma
  - Trustees of the University of Pennsylvania; Neurology, Philadelphia, Pennsylvania
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Maxine Mesinger MS Clinic/Baylor College of Medicine; Neurology, Houston, Texas
  - Neurological Associates, Inc., Richmond, Virginia
  - Swedish Neuroscience Institute; Multiple Sclerosis Center, Seattle, Washington
- Australia (2):
  - Royal Hobart Hospital, Hobart, Tasmania
  - St Vincent's Hospital Melbourne; Clinical Neuroscience and Neurological Research, Fitzroy, Victoria
- Austria (5):
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck; Department fuer Neurologie, Innsbruck
  - Kepler Universitätsklinikum GmbH - Neuromed Campus; Neurologie, Linz
  - Kepler Universitätskliniken GmbH - Med Campus III; Neurologie & Psychiatrie, Linz
  - Christian-Doppler-Klinik - Universitätsklinikum; Universitätskliniik für Neurologie, Salzburg
  - Medizinische Universitat Wien Medical University of Vienna, Vienna
- Belgium (2):
  - CHU Tivoli, La Louvière
  - AZ Alma vzw (Sijsele), Sijsele
- Brazil (4):
  - Hospital das Clinicas - UFG;Reumatologia, Goiânia, Goiás
  - Santa Casa de Misericordia; de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Universitario Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
- Bulgaria (2):
  - Shat Np Sveti Naum; 3Rd Clinic of Neurology, Sofia
  - Multiprofile Hosp. for Active Treatment;National Cardiology Hosp., Sofia
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - University of British Columbia UBC Hospital; Multiple Sclerosis (MS) Clinic - Vancouver, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Czechia (3):
  - Fakultni nemocnice Brno; Interni kardiologicka klinika, Brno
  - Vseobecna fakultni nemocnice v Praze; MS Centrum, Neurologicka klinika, Prague
  - Krajska zdravotni, a. s. ? Nemocnice Teplice, o. z.; Neurologicke oddeleni, Teplice
- Finland (3):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Tampereen yliopisto; Kliinisen lääketieteen laitos, Neurologian yksikkö, Tampere
  - Turku University Central Hospital; Pharmacy, Turku
- France (17):
  - Groupe Hospitalier Pellegrin; Service de neurochirurgie B, Bordeaux
  - Hopital Neurologique et Neurochirurgical Pierre Wertheimer; Service de Neurologie A, Bron
  - Hopital Cote De Nacre; Unite Neurologie Generale, Caen
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand; Service de Neurologie B, Clermont-Ferrand
  - Hopital Roger Salengro Service de Neurologie, Lille
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - CHRU Nancy; Service de neurologie, Nancy
  - Hôpital Guillaume et René Laënnec; Service Neurologie, Nantes
  - Hôpital Pasteur; Service de Neurologie, Nice
  - Groupe Hospitalo-Universitaire Caremeau; Service Neurologie, Nîmes
  - Fondation Rothschild; Service de Neurologie, Paris
  - Groupe Hospitalier Pitié- Salpétrière; Service Neurologie, Paris
  - Hôpital de Poissy; Service neurologie, Poissy
  - Hôpital Maison Blanche; Service de Neurologie, Reims
  - Chu De Strasbourg; Hopital Civil, Strasbourg
  - Hopital Purpan; Fédération de neurologie, Toulouse
- Germany (18):
  - Klinikum Bayreuth GmbH; Neurologische Klinik, Bayreuth
  - Marianne-Strauß-Klinik; Behandlung Kempfen für Multip Sklero Kranke gemeinnütz GmbH, Berg
  - Charite - Universitatsmedizin Berlin; Klinik fur Neurologie, Berlin
  - Jüdisches Krankenhaus Berlin; Abteilung fur Neurologie, Berlin
  - Berufsgenossenschaftliches Uni-Klinikum Bergmannsheil GmbH, Bochum
  - Kliniken der Stadt Koln gGmbH, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Neurologie, Dresden
  - Heinrich Heine Universität Düsseldorf; Neurologische Klinik, Düsseldorf
  - Klinikum Joh.Wolfg.Goethe-UNI Senckenbergisches Institut für Neuroonkologie, Frankfurt am Main
  - Universitätsklinikum Gießen und Marburg GmbH; Neurologie, Giessen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universität Leipzig; Innere Medizin, Neurologie, Dermatologie, Leipzig
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitatsklinikum Munster, Münster
  - Medizinische Einrichtungen des Bezirks Oberpfalz GmbH; Neurologie, Regensburg
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
  - DKD Helios Klinik (Deutsche Klinik für Diagnostik GmbH), Wiesbaden
- Greece (3):
  - 401 Military Hospital of Athens; Neurology Department, Athens
  - AHEPA Univ. General Hospital of Thessaloniki; B' Neurology Dept., Thessaloniki
  - Georgios Papanikolaou General Hosp. of Thessaloniki, Thessaloniki
- Hungary (6):
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Jahn Ferenc Del-Pesti Korhaz es Rendelointezet, Budapest
  - Vaszary Kolos Korhaz; Neurology, Esztergom
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ; Neurológiai Klinika, Szeged
  - Veszprém Megyei Csolnoky Ferenc Kórház; Reumatológia, Veszprém
- Israel (6):
  - Barzilai Medical Center; Neurology Department, Ashkelon
  - Hadassah University Hospital Ein Kerem; Neurology Department, Jerusalem
  - Rabin Medical Center; Multiple Sclerosis Clinic, Petah Tikva
  - The Chaim Sheba Medical Center; Multiple Sclerosis Center, Ramat Gan
  - Medical Center Ziv Safed; Neurology Department, Safed
  - Tel Aviv Sourasky Medical Center; Department of Neurology, Tel Aviv
- Italy (4):
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Hospital San Raffaele, Milan, Lombardy
  - Azienda Sanitaria Ospedaliera S. Luigi Gonzaga; Centro Regionale Sclerosi Multipla - Neurologia II, Orbassano, Piedmont
  - Ospedale Binaghi; Centro Sclerosi Multipla, Cagliari, Sardinia
- Lithuania (3):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital Public Institution, Klaipėda
  - Siauliai Hospital, Šiauliai
- Mexico (4):
  - Instituto Nacional de Neurologia y Neurocirugia, Mexico City, Mexico CITY (federal District)
  - Eleccion Salud SC, México, Mexico CITY (federal District)
  - Centro de Estudios Clinicos y Espec. Med. SC, Monterrey, Nuevo León
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
- Netherlands (2):
  - Erasmus MC; Afdeling Neurologie, Rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
- New Zealand (2):
  - Waikato Hospital; Neurology, Hamilton
  - Wellington Hospital; Department of Neurology, Wellington
- Oslo universitetssykehus HF, Ullevål; Nevrologisk avdeling, Oslo, Norway
- Peru (3):
  - Hospital IV Alberto Sabogal Sologuren; Unidad de Investigacion, Bellavista
  - Clinica Anglo Americana, Lima
  - Hospital Nacional Dos de Mayo - Centro de Investigacion en Oncología, Lima
- Poland (7):
  - Niepubliczny Zaklad Opieki Zdrowotnej KENDRON ; Poradnia Neurologiczna, Bialystok
  - Zespol Opieki Zdrowotnej w Konskich; Oddzial Neurologiczny, Gmina Końskie
  - Akson - Clinical Research Maciejowski - Bielecki Sp. Jawna, Jarosław
  - Diagnomed Clinical Research Sp. z o.o., Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej; Neuro-Medic, Katowice
  - SPZOZ Uni. Szpital Kliniczny nr 1 im. Norberta Barlickiego Uni. Medycznego w Lodzi ; Neurologii, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie; Klinika Neurochirurgii i Neurochirurgii Dzi, Lublin
- Portugal (6):
  - Hospital Garcia de Orta; Servico de Neurologia, Almada
  - Hospital Prof. Dr. Fernando Fonseca; Servico de Neurologia, Amadora
  - HUC; Servico de Neurologia, Coimbra
  - Hospital Geral; Servico de Neurologia, Coimbra
  - Hospital de Santa Maria; Servico de Neurologia, Lisbon
  - Hospital Geral de Santo Antonio; Servico de Neurologia, Porto
- Romania (4):
  - Elias Emergency University Hospital Neurology Dept; Neurology Department, Bucharest
  - SC Clubul Sanatatii SRL, Campulung Muscel
  - Spitalul Clinic Judetean de Urgenta Targu Mures; Clinica Neurologie, Târgu Mureş
  - Timisoara Emergency County Clinical Hospital, Timi?oara
- Research Medical Complex "Vashe Zdorovie"; Neurology Department, Kazan', Tatarstan Republic, Russia
- Spain (14):
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Neurologia, Salt, Girona
  - Hospital Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Intermedios y Urgencias Pediatricas, Santiago de Compostela, LA Coruña
  - Hospital de Basurto Servicio de Neurologia, Bilbao, Vizcaya
  - Hospital General Univ. de Alicante, Alicante
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Neumo-Inmunologia, Barcelona
  - Hospital Clinic i Provincial; Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Universitario de La Princesa; Servicio de Neurología, Madrid
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Neurología, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Neurologia, Málaga
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
- Switzerland (2):
  - Universitätsspital Basel; Neurologie, Basel
  - Ospedale Regionale di Lugano - Civico; Neurologia, Lugano
- Ukraine (11):
  - CNPE City Clinical Hospital #3 of Chernivtsi City Council, Chernivtsi, Chernihiv Governorate
  - Municipal Non-profit Enterprise Odessa Regional Clinical Hospital of Odessa Regional Council, Odesa, Kherson Governorate
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, KIEV Governorate
  - Ukrainian State Inst. of Med. and Social Problems of Disability; Neuro, Dnipropetrovsk
  - Dnipropetrovsk State Medical Academy; Dept of Neurology, Dnipropetrovsk
  - Ams of Ukraine; Inst. of Neurology, Psychiatry & Narcology, Kharkiv
  - Kh. Med. Ac. of P.-Gr. Ed.; Cl. Cen. Hosp. of UkrZal.; 3rd Dept. Neurology, Kharkiv
  - Kyiv City Clinical Hospital #4 MAHC of Kyiv; Chair of Neurology, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Clinical Hospital; Department of Neurology, Lviv
  - Vinnytsya National Med. Uni. n.a. M.I. Pyrohov; Dept. of Neurology #3, Vinnytsia
- United Kingdom (5):
  - Walton Centre NHS Foundation Trust, Neuroscience Research Centre; CLINICAL TRIALS UNIT, Liverpool
  - Barts and the London NHS Trust, London
  - Kings College Hospital; Neurology, London
  - Royal Victoria Infirmary; Neurology Dept., Newcastle upon Tyne
  - Uni Hospital Queens Medical Centre; Neurology, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203
- [Derived] Zivadinov R, Pei J, Clayton D, Goldman DE, Winger RC, Cabatingan MS, Dwyer MG, Bergsland N. Evolution of atrophied T2 lesion volume in primary-progressive multiple sclerosis: results from the phase 3 ORATORIO study. J Neurol Neurosurg Psychiatry. 2024 May 14;95(6):536-543. doi: 10.1136/jnnp-2023-332573. PMID 38071574
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Hauser SL, Bar-Or A, Weber MS, Kletzl H, Gunther A, Manfrini M, Model F, Mercier F, Petry C, Wing Q, Koendgen H, Smith T, Kappos L. Association of Higher Ocrelizumab Exposure With Reduced Disability Progression in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2023 Feb 15;10(2):e200094. doi: 10.1212/NXI.0000000000200094. Print 2023 Mar. PMID 36792367
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Arnold DL, Sprenger T, Bar-Or A, Wolinsky JS, Kappos L, Kolind S, Bonati U, Magon S, van Beek J, Koendgen H, Bortolami O, Bernasconi C, Gaetano L, Traboulsee A. Ocrelizumab reduces thalamic volume loss in patients with RMS and PPMS. Mult Scler. 2022 Oct;28(12):1927-1936. doi: 10.1177/13524585221097561. Epub 2022 Jun 7. PMID 35672926
- [Derived] Butzkueven H, Spelman T, Horakova D, Hughes S, Solaro C, Izquierdo G, Kubala Havrdova E, Grand'Maison F, Prat A, Girard M, Hupperts R, Onofrj M, Lugaresi A, Taylor B; MSBase Study Group; Giovannoni G, Kappos L, Hauser SL, Montalban X, Craveiro L, Freitas R, Model F, Overell J, Muros-Le Rouzic E, Sauter A, Wang Q, Wormser D, Wolinsky JS. Risk of requiring a wheelchair in primary progressive multiple sclerosis: Data from the ORATORIO trial and the MSBase registry. Eur J Neurol. 2022 Apr;29(4):1082-1090. doi: 10.1111/ene.14824. Epub 2021 May 6. PMID 33724638
- [Derived] Wolinsky JS, Arnold DL, Brochet B, Hartung HP, Montalban X, Naismith RT, Manfrini M, Overell J, Koendgen H, Sauter A, Bennett I, Hubeaux S, Kappos L, Hauser SL. Long-term follow-up from the ORATORIO trial of ocrelizumab for primary progressive multiple sclerosis: a post-hoc analysis from the ongoing open-label extension of the randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2020 Dec;19(12):998-1009. doi: 10.1016/S1474-4422(20)30342-2. Epub 2020 Oct 29. PMID 33129442
- [Derived] Fox EJ, Markowitz C, Applebee A, Montalban X, Wolinsky JS, Belachew S, Fiore D, Pei J, Musch B, Giovannoni G. Ocrelizumab reduces progression of upper extremity impairment in patients with primary progressive multiple sclerosis: Findings from the phase III randomized ORATORIO trial. Mult Scler. 2018 Dec;24(14):1862-1870. doi: 10.1177/1352458518808189. Epub 2018 Nov 12. PMID 30415593
- [Derived] Wolinsky JS, Montalban X, Hauser SL, Giovannoni G, Vermersch P, Bernasconi C, Deol-Bhullar G, Garren H, Chin P, Belachew S, Kappos L. Evaluation of no evidence of progression or active disease (NEPAD) in patients with primary progressive multiple sclerosis in the ORATORIO trial. Ann Neurol. 2018 Oct;84(4):527-536. doi: 10.1002/ana.25313. PMID 30155979
- [Derived] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 943 participants were screened and 732 were randomized into the study, of which 725 received at least one dose of placebo or ocrelizumab.
Period: Overall Study
Arm/Group | Placebo | Ocrelizumab 600 mg
Started | 244 | 488
Completed | 89 | 218
Not Completed | 155 | 270
Not completed — Adverse Event | 22 | 40
Not completed — Death | 6 | 20
Not completed — Lack of Efficacy | 32 | 33
Not completed — Lost to Follow-up | 4 | 15
Not completed — Non-Compliance | 2 | 2
Not completed — Non-Compliance With Study Drug | 2 | 2
Not completed — Other | 18 | 47
Not completed — Physician Decision | 10 | 25
Not completed — Protocol Violation | 1 | 2
Not completed — Study Terminated By Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 57 | 82
Not completed — Pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) population which included all randomized participants in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ocrelizumab 600 mg | Total
Number analyzed (Participants) | 244 | 488 | 732
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 244 | 488 | 732
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (8.3) | 44.7 (7.9) | 44.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 237 | 361
  Male | 120 | 251 | 371
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 32 | 46
  Not Hispanic or Latino | 206 | 385 | 591
  Unknown or Not Reported | 24 | 71 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 5 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 235 | 454 | 689
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 20 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Clinical Disability Progression (CDP) Sustained for at Least 12 Weeks During the Double-Blind Treatment Period
Description: The time to onset of CDP was defined as time from baseline to first disability progression, which is confirmed at next regularly scheduled visit >=12 weeks (>=84 days) after initial disability progression. Baseline for time to onset of CDP is the date of randomization, independent of the first day of dosing. Disability progression is defined as an increase of >= 1.0 point from baseline expanded disability status scale (EDSS) score, if baseline EDSS value is <=5.5 points (inclusive), or an increase of >=0.5 points, if baseline EDSS is >5.5 points. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). The randomized participants who did not receive any treatment were censored at days 0 in each Arm.
Time Frame: Maximal follow up: 216 weeks for Placebo arm and 217 weeks for Ocrelizumab arm
Population: ITT population included all randomized participants in the study. Number of participants analyzed is the total participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 244 | 487
weeks | NA [0 to NA] — The median and upper limit of full range for time to onset of CDP has not been reached due to low number of participants with the event at the end of the study. | NA [0 to NA] — The median and upper limit of full range for time to onset of CDP has not been reached due to low number of participants with the event at the end of the study.

2. Secondary Outcome: Time to Onset of Clinical Disability Progression (CDP) Sustained for at Least 24 Weeks During the Double-Blind Treatment Period
Description: as for outcome 1
Time Frame: Maximal follow up: 216 weeks for Placebo arm and 217 weeks for Ocrelizumab arm
Population: ITT population included all randomized participants in the study. Number of participants analyzed is the total participants who were evaluable for this endpoint.
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 244 | 487
weeks | NA [0 to NA] — The median and upper limit of full range for time to onset of CDP has not been reached due to low number of participants with the event at the end of the study. | NA [0 to NA] — The median and upper limit of full range for time to onset of CDP has not been reached due to low number of participants with the event at the end of the study.

3. Secondary Outcome: Percent Change From Baseline in Timed 25-Foot Walk (T25-FW) at Week 120
Time Frame: Baseline, Week 120
Population: ITT population included all randomized participants in the study. Here, number of participants analyzed is the total participants who were evaluated for this endpoint. Here, least square mean is indicating adjusted geometric mean.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 239 | 473
percent change | 55.097 [39.855 to 71.999] | 38.933 [29.222 to 49.374]
Statistical Analysis 1: Comparison: Placebo vs Ocrelizumab 600 mg; Estimates (back-transformed) based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix: log(Post-baseline(BL)/BL) = log(BL 25-FTW) + Geographical Region (US vs. ROW) + Age (<=45, > 45 years) + Week + Treatment + Treatment*Week (repeated values over Week) + log (BL 25-FTW)*Week. Relative reduction was calculated as -Relative change = -(OCR response-Placebo response)/Placebo response*100%. The 95% CI for relative reduction was obtained using the Bootstrap method; Test type: Superiority or Other; p = 0.0404, Ranked ANCOVA — P-value from a ranked ANCOVA on Percent Change from BL adjusting for rank of BL 25-Foot Timed Walk (25-FTW), Geographical Region (US vs ROW) and Age (<=45, > 45 years); missing observations imputed with LOCF; Relative Reduction (%) = 29.337, 95% CI 2-sided [-1.618 to 51.456] — Relative reduction was calculated as -Relative change = - (Ocrelizumab response-Placebo response)/Placebo response*100%. The 95% CI for relative reduction was obtained using the Bootstrap method

4. Secondary Outcome: Percent Change From Baseline in Total Volume of T2 Lesions at Week 120
Time Frame: From Baseline to Week 120
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 234 | 464
percent change | 7.426 [4.967 to 9.942] | -3.366 [-4.987 to -1.718]
Statistical Analysis 1: Comparison: Placebo vs Ocrelizumab 600 mg; Estimates (back-transformed) are based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix: log(Post-BL/BL) = log(BL T2 lesion volume) + Geographical Region (US vs. ROW) + Age (<=45, > 45 years) + Week + Treatment + Treatment*Week (repeated values over Week) + log (BL T2 lesion volume)*Week; Test type: Superiority or Other; p < 0.0001, Ranked ANCOVA — P-value is from ranked ANCOVA on Percent Change from BL adjusting for rank of BL T2 lesion volume, Geographical Region (US vs ROW) and Age (<=45, > 45 years); missing observations imputed with LOCF; Ratio of Adjusted Geometric Means = 0.9, 95% CI 2-sided [0.876 to 0.924]

5. Secondary Outcome: Percent Change in Total Brain Volume From Week 24 to Week 120
Time Frame: From Week 24 to Week 120
Population: ITT population included all randomized participants in the study. Number of participants analyzed is the total participants who were evaluable for this endpoint. Here, least square mean is indicating adjusted mean.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 203 | 407
percent change | -1.093 [-1.236 to -0.951] | -0.902 [-1.004 to -0.799]
Statistical Analysis 1: Comparison: Placebo vs Ocrelizumab 600 mg; Estimates are from analysis based on MMRM using unstructured covariance matrix: Percentage Change = Brain Volume at Week 24 + Geographical Region (US vs. ROW) + Age (<=45, > 45 years) + Week + Treatment + Treatment*Week (repeated values over Week) + Brain Volume at Week 24*Week. Relative reduction was calculated as - Relative change = - (OCR response-Placebo response)/Placebo response*100%. The 95% CI for relative reduction was obtained using Bootstrap method; Test type: Superiority or Other; p = 0.0206, MMRM; Relative Reduction (%) = 17.475, 95% CI 2-sided [3.206 to 29.251] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change in From Baseline Physical Component Summary Score (PCS) SF- 36 Health Survey (SF-36) at Week 120
Description: The SF-36v2 is a 36-item, self- reported, generic measure of quality of life that has been widely used in multiple disease areas. It is composed of 8 health domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The PCS score was derived based on the SF-36 V2 User's Manual. Scoring for PCS involves (a) recoding item response values, (b) summing recoded response values for all items in a given scale to obtain the scale raw score, (c) transforming scale raw score to a 0-100 score. The PCS score was computed by (a) multiplying each health domain z score by a scale-specific physical factor score coefficient, (b) summing the resulting products, (c) converting the product total to T score. The total score ranges from 0-100, higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: From Baseline to Week 120
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Ocrelizumab 600 mg
Number analyzed (Participants) | 128 | 292
units on a scale | -1.108 [-2.394 to 0.177] | -0.731 [-1.655 to 0.193]
Statistical Analysis 1: Comparison: Placebo vs Ocrelizumab 600 mg; Estimates are from analysis based on MMRM using unstructured covariance matrix: Change = Baseline PCS Score + Geographical Region (US vs. ROW) + Age (<=45, > 45 years) + Week + Treatment + Treatment*Week (repeated values over Week) + Baseline PCS Score*Week; Test type: Superiority or Other; p = 0.6034, MMRM; Difference in Adjusted Means = 0.377, 95% CI 2-sided [-1.048 to 1.802], Standard Error of Mean 0.725 — Difference in adjusted mean was calculated as Ocrelizumab SF-36 Physical Component Summary Score - Placebo SF-36 Physical Component Summary Score

7. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: AEs included infusion related reactions (IRRs) and serious multiple sclerosis (MS) relapses, but excluded non-serious MS relapses.
Time Frame: From baseline to 9 years
Population: The safety population includes all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Placebo (Open Label Extension); Ocrelizumab (Open Label Extension): During the OLE phase, all participants received ocrelizumab 600-mg IV infusion every 24 weeks.
Arm/Group | Placebo | Ocrelizumab 600 mg | Placebo (Open Label Extension) | Ocrelizumab (Open Label Extension)
Number analyzed (Participants) | 239 | 486 | 158 | 369
Participants
  Serious Adverse Events | 53 | 99 | 59 | 167
  Adverse Events | 215 | 462 | 148 | 354

ADVERSE EVENTS:
Time Frame: Baseline up to 615 weeks
Description: The safety population included all participants who received any study drug.
Arm/Group | DB PLACEBO | DB OCRELIZUMAB | OLE PLACEBO | OLE OCRELIZUMAB
All-Cause Mortality (participants affected / at risk) | 3/239 | 3/486 | 4/158 | 19/369
Serious Adverse Events (participants affected / at risk) | 58/239 | 104/486 | 59/158 | 167/369
Other Adverse Events (participants affected / at risk) | 175/239 | 400/486 | 134/158 | 318/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB PLACEBO (N=239) | DB OCRELIZUMAB (N=486) | OLE PLACEBO (N=158) | OLE OCRELIZUMAB (N=369)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
EPIRETINAL MEMBRANE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE INFLAMMATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETINAL DISORDER (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAL POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANORECTAL VARICES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL POLYP HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
CATHETER SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRUG INTOLERANCE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTHERMIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABSCESS OF EYELID (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
APPENDICITIS PERFORATED (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BORRELIA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CANDIDA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 3 (3) | 2 (6) | 5 (8)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 12 (12)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 31 (31)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DENGUE FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HEPATITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES OPHTHALMIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LARGE INTESTINE INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MASTITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MENINGITIS ASEPTIC (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (4) | 6 (7) | 3 (4) | 17 (18)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELOCYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 7 (10)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUSPECTED COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 4 (4) | 7 (10) | 20 (28)
UROSEPSIS (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 7 (7)
VESTIBULAR NEURONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VIRAL PERICARDITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ZIKA VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
CARDIAC CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
INCISION SITE IMPAIRED HEALING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL FEVER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD GLUCOSE FLUCTUATION (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HELICOBACTER TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SERONEGATIVE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPLASTIC LARGE-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BENIGN PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BENIGN VAGINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BORDERLINE SEROUS TUMOUR OF OVARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
CHONDROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRADUCTAL PAPILLARY BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT FIBROUS HISTIOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NODULAR MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PARAGANGLION NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ROSAI-DORFMAN SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
EMBOLIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
MULTIPLE SCLEROSIS PSEUDO RELAPSE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
MUSCLE SPASTICITY (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRIMARY PROGRESSIVE MULTIPLE SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (7)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 2 (4) | 2 (3) | 2 (5)
UHTHOFF'S PHENOMENON (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BEHAVIOUR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BLADDER PERFORATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERMENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST TORSION (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HYPERSENSITIVITY PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD THICKENING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
DRY GANGRENE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB PLACEBO (N=239) | DB OCRELIZUMAB (N=486) | OLE PLACEBO (N=158) | OLE OCRELIZUMAB (N=369)
CONSTIPATION (Gastrointestinal disorders) | 12 (14) | 25 (28) | 8 (8) | 23 (23)
DIARRHOEA (Gastrointestinal disorders) | 12 (15) | 27 (43) | 11 (15) | 42 (54)
FATIGUE (General disorders) | 24 (32) | 30 (33) | 12 (14) | 24 (30)
BRONCHITIS (Infections and infestations) | 15 (21) | 30 (40) | 11 (15) | 32 (52)
INFLUENZA (Infections and infestations) | 21 (25) | 57 (76) | 16 (21) | 39 (59)
NASOPHARYNGITIS (Infections and infestations) | 63 (125) | 117 (206) | 48 (95) | 100 (190)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 (21) | 60 (87) | 14 (17) | 56 (110)
URINARY TRACT INFECTION (Infections and infestations) | 57 (117) | 103 (255) | 44 (120) | 127 (488)
CONTUSION (Injury, poisoning and procedural complications) | 19 (22) | 14 (19) | 9 (13) | 23 (35)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 61 (154) | 194 (496) | 40 (98) | 56 (178)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 30 (39) | 56 (66) | 23 (36) | 57 (73)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 38 (54) | 59 (71) | 23 (30) | 54 (70)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25 (31) | 35 (38) | 18 (23) | 33 (38)
DIZZINESS (Nervous system disorders) | 10 (12) | 27 (33) | 10 (13) | 14 (17)
HEADACHE (Nervous system disorders) | 31 (48) | 68 (98) | 15 (19) | 41 (73)
DEPRESSION (Psychiatric disorders) | 31 (35) | 34 (35) | 9 (9) | 23 (24)
INSOMNIA (Psychiatric disorders) | 15 (15) | 28 (31) | 10 (10) | 12 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 35 (44) | 12 (13) | 38 (45)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 10 (11) | 21 (26)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 10 (13) | 25 (36)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 11 (12) | 22 (25)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 14 (23) | 23 (39)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 21 (22) | 76 (87)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 21 (22) | 76 (87)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 6 (10) | 20 (26)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 20 (38)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 16 (28) | 40 (75)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 8 (8) | 12 (14)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 19 (21)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 9 (14) | 8 (18)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8) | 14 (17)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 23 (24)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 12 (12) | 28 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT01194570/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT01194570/SAP_001.pdf